CLINICAL TRIAL: NCT01672554
Title: Open Label, Non-randomised, Single Arm, Phase IIIB Switch Study: Evaluating the Clinical Benefits of Quetiapine XR in Patients With Schizophrenia and Anxiety Disorder.
Brief Title: Clinical Benefits of Seroquel XR in Anxiety Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Corporation de Recherche en Neuropsycho Pharmacologie de Quebec (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443C00030
Record Dates: First submitted 2012-08-20; First posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Schizophrenia; Anxiety
Keywords: Schizophrenia; Anxiety disorder
MeSH Terms: conditions — Schizophrenia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seroquel XR (Other): Quetiapine XR will be titrated according to the following pattern: Seroquel XR 300 mg on day 1 and Seroquel XR 600 mg on day 2. On day 3, the dosage could be either maintained at 600 mg/day or continued up to 800 mg/day or if the 600 mg dose is not tolerated, the dose could then be reduced to 400 mg/day. Following this, subjects will be flexibly dosed, according to clinical judgment of the investigator, between 400 mg/day and 800 mg/day with minimum dose adjustments of 200 mg/day. This adjustment can be performed at anytime during the study but should not take place within a week from last cognitive assessment, planned at month 6. An overlap of at least 4 days but not more than 2 weeks with the previous antipsychotic will be allowed with decreasing doses on a two-week period.
  Interventions: Drug: Quetiapine XR

INTERVENTIONS:
Drug: Quetiapine XR — Quetiapine XR will be titrated according to the following pattern: Seroquel XR 300 mg on day 1 and Seroquel XR 600 mg on day 2. On day 3, the dosage could be either maintained at 600 mg/day or continued up to 800 mg/day or if the 600 mg dose is not tolerated, the dose could then be reduced to 400 mg/day. Following this, subjects will be flexibly dosed, according to clinical judgment of the investigator, between 400 mg/day and 800 mg/day with minimum dose adjustments of 200 mg/day. This adjustment can be performed at anytime during the study but should not take place within a week from last cognitive assessment, planned at month 6. An overlap of at least 4 days but not more than 2 weeks with the previous antipsychotic will be allowed with decreasing doses on a two-week period.

SUMMARY:
This research will explore whether Quetiapine XR used primarily to treat psychosis may also cover for comorbid anxiety disorder and offer advantages in patients with schizophrenia and comorboid anxiety disorder. Preliminary data on pharmacological properties of Quetiapine and its metabolites and intuitive impression from our clinical experience lead to believe that Seroquel XR use in monotherapy may offer advantages over other antipsychotics in treating co-morbid anxiety disorder in patients suffering from schizophrenia. This open label switch study conducted in a schizophrenic population intends to verify this hypothesis.

DETAILED DESCRIPTION:
This is an open label, non-randomised, single arm phase IIIB study. Patients will be enrolled in this study if their current antipsychotic medication does not provide optimal control of psychopathology symptoms, as judged by the investigator. Therefore, the patients will not be switched from their current effective and well tolerated antipsychotic regimen to the study drug for the sole reason of being enrolled into the study. After enrolment, patients will be switched to Quetiapine XR and followed in an intent-to-treat design over 6 months. Even if a patient should stop for any reason Quetiapine XR or require adding or adjusting an antidepressant for anxiety resistant symptoms, he/she will be assessed for the entire study. Data will be analysed separately.

Quetiapine XR will be titrated according to the following pattern: Seroquel XR 300 mg on day 1 and Seroquel XR 600 mg on day 2. On day 3, the dosage could be either maintained at 600 mg/day or continued up to 800 mg/day or if the 600 mg dose is not tolerated, the dose could then be reduced to 400 mg/day. Following this, subjects will be flexibly dosed, according to clinical judgment of the investigator, between 400 mg/day and 800 mg/day with minimum dose adjustments of 200 mg/day. This adjustment can be performed at anytime during the study but should not take place within a week from last cognitive assessment, planned at month 6. An overlap of at least 4 days but not more than 2 weeks with the previous antipsychotic will be allowed with decreasing doses on a two-week period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent;
* A diagnosis of schizophrenia or schizophrenia spectrum psychosis (schizophreniform, schizoaffective, delusional disorder, brief psychosis) as defined by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV);
* Presenting a co-morbid anxiety disorder not well controlled with the current pharmacological treatment according to the investigator corresponding to DSM-IV;
* Having an initial score of more than 20 at enrolment on HAM-A scale;
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment;

Exclusion Criteria:

* Patient with an antidepressant or benzodiazepine recently (last 4 weeks) introduced, or that had requested a dosing adjustment in the last 4 weeks;
* Patient with an anticholinergic taken on a regular basis;
* Patient receiving more than one antipsychotic;
* Pregnancy or lactation;
* Any DSM-IV Axis I disorder not defined in the inclusion criteria;
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others;
* Known intolerance or lack of response to Quetiapine fumarate, as judged by the investigator;
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir;
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids;
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before enrolment;
* Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria;
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment;
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment;
* Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator;
* Involvement in the planning and conduct of the study;
* Previous enrolment of treatment in the present study;
* Participation in a phase I-II-III drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements;
* A patient with Diabetes Mellitus (DM) - An absolute neutrophil count (ANC) of 1.5 x 109 per liter;
* An ALT-AST count of 3 x ULN and/or Bilirubin count 1.5 x ULN;
* Any clinically significant laboratory abnormality, as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-04 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Anxiety disorder | Clinical anxiety scales will be assessed over 6 months at the following visits: day 1, day 7, day 14, month 1, month 2, month 3 and month 6.
  Our main objective will be to assess over 6 months, the impact of a switch to Seroquel XR in subjects suffering from schizophrenia associated with a co morbid anxiety disorder as measured by well-validated clinical anxiety scales.

SECONDARY OUTCOMES:
Tolerability and safety | Evaluated at each visit over 6 months: day 1, day 7, day 14, month 1, month 2, month 3 and month 6.
  To assess tolerability and safety profile after a switch to Seroquel XR in such population over 6 months. To do so a pharmacological evaluation will collected, this includes spontaneous patient self-report of any adverse event. The UKU (Udvalg for klinedke Undersodgelser)side effect rating scale will also address drug side effects. The patient perception of medication will be assessed by the Drug Attitude Inventory (DAI) scale and will be used as a compliance indicator. Extrapyramidal Symptom Rating Scale (ESRS) will be performed to assess extrapyramidal side effects. Current concomitant medication will be recorded also.

OTHER OUTCOMES:
Cognition | The Matrics consensus battery will be performed at the baseline visit and at the end of study visit.
  To assess cognitive performance after a switch to Seroquel XR in such population over 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roch-Hugo Bouchard, MD, FRCPC, Principal Investigator — Laval University
Locations (1):
- CRNPQ, Québec, Quebec, Canada